CLINICAL TRIAL: NCT04387240
Title: Evaluating the Efficacy of Artesunate in Adults With Mild Symptoms of COVID-19
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: did not get enough fund and IRB request
Sponsor: Princess Nourah Bint Abdulrahman University (Other)
Responsible Party: Principal Investigator, osama y kentab, Clinical Associate Professor of Emergency Medicine, Princess Nourah Bint Abdulrahman University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20-0192
Record Dates: First submitted 2020-05-12; First posted 2020-05-13 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Covid 19 Positive; Corona Virus Infection
Keywords: artemisinin; Artesunate
MeSH Terms: conditions — Coronavirus Infections | interventions — artemisinin; Artesunate

STUDY DESIGN:
Intervention Model Description: double blind controlled trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: the pharmacy will do the randomization of the labeled drug and placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): this group will receive the Artemisinin / Artesunate 100mg once daily for 5 days
  Interventions: Drug: Artemisinin / Artesunate
- placibo (Placebo Comparator): this group will receive a placebo of the same shape and picture of the study drug
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Artemisinin / Artesunate — testing the drug capabilities in reducing the shedding and causing the testing for covid 19 to become negative
  Arms: intervention group
Other: placebo — placebo or sham drug will be given to the second arm
  Arms: placibo

SUMMARY:
Coronavirus disease (COVID-19) is an infectious disease caused by a newly discovered coronavirus.

At this time, there are no specific vaccines or treatments for COVID-19. However, there are many ongoing clinical trials evaluating potential treatments Drugs used to treat malaria infection has shown to be beneficial for many other diseases, including viral infections.

In this Clinical trial, Investigators will evaluate the effect of Artemisinin / Artesunate on morbidity of COVID-19 patients in decreasing the course of the disease and viral load in symptomatic stable positive swab COVID-19 patients. Investigators are hypothesizing that due to the antiviral properties of this drug it will help as a treatment for the COVID -19 patients. In improving their condition and clearing the virus load,

DETAILED DESCRIPTION:
In this Clinical trial, Investigators will evaluate the effect of Artemisinin / Artesunate on morbidity of COVID-19 patients in decreasing the course of the disease and viral load in symptomatic stable positive swab COVID-19 patients. investigators are hypothesizing that due to the antiviral properties of this drug it will help as a treatment for the COVID -19 patients. In improving their condition and clearing the virus load, investigators are testing two groups the one that will take the drug and then compare them to a placebo group that will not take any drug for the treatment in a blinded fashion made by randomization done by our pharmacy team so investigators eliminate risk of bias. Our expectation is to find a total reduction of the hospital stay to 7 days instead of 14 days currently indicating the effectiveness of the medication in eradicating the virus.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient age more than 18 and less than 60 years
* Symptomatic , positive swab covid-19 patients
* Patients who have mild to moderate symptoms
* Patients who have no risk factors like
* Patients who is not on other medications rather those on supportive care

Exclusion Criteria:

* · Patients who have sever disease- shortness of breath, sick patients or admitted in ICU

  * Patients who are receiving ventilation supports
  * High risk group like :- age more than 60 years, chronic heart diseases, chronic lungs diseases, diabetes, immunocompromised diseases or on immune suppression medications or pregnant women
  * Patients who are on other medications which used as treatment for covid 19

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
length of stay in hospital | within the first 6 days intervention
  absence of the virus shedding evidenced by negative swabs

SECONDARY OUTCOMES:
number of ICU admission | 14 days
  reduction of morbidity and mortality
resolution of symptoms | 6 days - 10 day
  finding the time that the symptoms disappear

CONTACTS AND LOCATIONS:
Overall Officials: Osama Kentab, MD, Principal Investigator — Princess Nourah Bint Abdulrahman University
Locations (1):
- Princess Nourah Bint Abdulrahman Univeristy, Riyadh, Central, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No